CLINICAL TRIAL: NCT02987998
Title: A Phase I Safety and Feasibility Study of Neoadjuvant Chemoradiation Plus Pembrolizumab Followed By Consolidation Pembrolizumab in Resectable Stage 3A Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant Chemoradiation Plus Pembrolizumab Followed By Consolidation Pembrolizumab in NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: higher than expected rate of toxicity & unrealistic timeline to complete trial under company's proposed plan to reopen
Sponsor: Nathan Pennell, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Nathan Pennell, MD, PhD, Study principal investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4516
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Stage IIIA Non-Small Cell Lung Cancer
Keywords: Pembrolizumab; Chemoradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; pembrolizumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Resectable Patients (Experimental): Chemoradiation (Cisplatin + Etoposide + Pembrolizumab with concurrent radiation). Patients will be assessed for surgery followed by consolidation therapy
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Pembrolizumab; Drug: Radiation

INTERVENTIONS:
Drug: Cisplatin — Cisplatin (50mg/m2 IV D1, 8, 29, 36)
Drug: Etoposide — Etoposide (50mg/m2 IV D1-5, 29-33)
Drug: Pembrolizumab — Pembrolizumab (200mg IV D1, 21, 42)
Drug: Radiation — Radiation (1.8Gy/D to 45Gy in 25 fractions)

SUMMARY:
The purpose of this study is to determine the feasibility and evaluate the safety of delivering chemoradiotherapy, the usual approach to non-small cell lung cancer, in combination with pembrolizumab (MK-3745), followed by consolidation pembrolizumab after surgical resection. Consolidation therapy is treatment given following the initial treatment.

Pembrolizumab is an investigational drug (also known as Keytruda), which has been approved by the FDA for use in certain types of skin cancer (melanoma), and for use in certain types of head and neck cancer. However, it has not been approved for use in other cancers such as non-small cell lung cancer (NSCLC). Pembrolizumab is a monoclonal antibody that binds to the surface of some cells of the immune system and activates them against cancer cells. It is not chemotherapy.

DETAILED DESCRIPTION:
The primary hypothesis is that the addition of pembrolizumab to neoadjuvant concurrent chemoradiation, followed by consolidation pembrolizumab, will be safe and feasible to deliver to patients with resectable stage 3A Non-small cell lung cancer (NSCLC).

This study also plans to observe the efficacy of this combination in the overall and biomarker-positive population.

Primary Objective Primary objective of this phase 1 study is to determine safety and feasibility of MK3475 with standard of care therapy of chemotherapy with radiation for newly diagnosed stage 3 lung carcinoma.

• To define the Safety, tolerability and feasibility of MK3475 in combination with chemotherapy with cisplatin and etoposide along with 45 Gy of radiation in newly diagnosed stage 3 non-small cell lung carcinoma.

Secondary Objective(s)

* Progression Free Survival
* Objective response rate,
* Complete pathologic response rate,
* Nodal downstaging at surgery,
* Overall survival,
* Safety and tolerability

Correlative Objective(s) Exploratory objectives: Overall response rate, progression free survival, overall survival in Programmed death-ligand (PDL-1) positive versus negative subgroups

Study Design This is an open-label, single arm phase I trial of neoadjuvant chemotherapy + pembrolizumab with concurrent radiation followed by surgical resection and consolidation pembrolizumab in resectable stage 3A (N2+) NSCLC.

Eligible patients will have biopsy-confirmed T1-3N2M0 (stage IIIA) non-small cell lung cancer (adenocarcinoma, squamous cell carcinoma, or large cell/NSCLC not otherwise specified), performance status 0-1, adequate lung function and deemed medically resectable by a thoracic surgeon, adequate organ function for chemotherapy, and no contraindications to pembrolizumab (i.e. autoimmune disorders or underlying pulmonary fibrosis).

Because pembrolizumab has been safely added to multiple platinum doublet chemotherapy regimens in lung cancer but not yet tested in the setting of concurrent radiation, we plan to evaluate safety and feasibility of the combination therapy. 10 patients will be enrolled at the full starting dose of all 3 agents. If 3 or more (>30%) have grade 3 or higher pulmonary toxicity or any grade 4 nonhematologic toxicity, the study will be stopped. If 2 or fewer have > grade 3 pulmonary toxicity or > grade 4 other nonhematologic toxicity, then an additional 10 will be enrolled. If 5 or fewer (<25%) of the 20 patients have > grade 3 pulmonary toxicity or > grade 4 other nonhematologic toxicity, then this regimen will be deemed safe and feasible for further study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage 3A Non-Small Cell Lung Cancer
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable or unmeasurable disease based on RECIST 1.1.
* Be willing to provide archival tissue from a tumor lesion or obtain a new biopsy if tissue unavailable.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology group (ECOG) Performance Scale.
* Demonstrate adequate organ function

  * Absolute neutrophil count (ANC) ≥1,500/mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or erythropoiesis dependency
  * Serum creatinine or Measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) or ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Serum total bilirubin ≤ 1.5 X ULN, or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * Aspartate transaminase (AST) (SGOT) and Alanine transaminase (ALT) (SGPT) ≤ 2.5 X ULN or ≤ 5 X ULN for subjects with liver metastases
  * Albumin ≥2.5 mg/dL
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had any prior chemotherapy, targeted small molecule therapy, or radiation therapy for the currently diagnosed cancer.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with grade 3 pulmonary toxicity or grade 4 other non hematologic toxicity | Up to 5 years
  If 5 or fewer (<25%) of the 20 patients have > grade 3 pulmonary toxicity or > grade 4 other nonhematologic toxicity, then this regimen will be deemed safe and feasible for further study

SECONDARY OUTCOMES:
Progression Free Survival | Up to 5 years
  Time from beginning of treatment to progression, death, or five years, whichever came first. Progression is defined as Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm
Objective Response Rate | Up to 5 years
  Number of patients with objective response (CR + PR) where complete response is defined as Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. And Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Complete Pathologic Response Rate | Up to 5 years
  Pathological complete response is defined as absence of foci of tumor cells at the local site (pCR)
Nodal Downstaging at Surgery | Up to 4 weeks after induction treatment
  Number of patients with reduced stages in nodes at surgery
Overall Survival | Up to 5 years
  Time from beginning of treatment to death or 5 year, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States